CLINICAL TRIAL: NCT06017700
Title: School-based Group Interpersonal Therapy for Adolescents With Depression in Nepal: a Pilot Realist Cluster-randomised Controlled Trial
Brief Title: School-based IPT-G for Adolescents With Depression in Nepal: a Pilot Realist C-RCT
Acronym: SAATHI-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Transcultural Psychosocial Organization Nepal (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MR/W00285X/1
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The study design is a parallel two-arm realist pilot cluster-randomised controlled trial. The trial will be conducted in eight schools (four intervention and four control). We will assess participants in intervention and control arms at baseline (week 0), after the first group session (week 5), after the sixth group session (week 12), at endline (weeks 20-21) and at follow-up (weeks 45-46). A caregiver survey will be administered at baseline and endline. Focus groups and interviews will be conducted with patients, caregivers, teachers, nurses, school principals.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPT-G (Experimental): Participants in the intervention arm will receive group interpersonal therapy in schools facilitated by trained laypersons. Groups are gender specific and comprise 6-8 adolescents. There are ten group sessions (approximately 90 min each, delivered weekly): in the first session the facilitator will focus on encouraging participants to review and share their interpersonal problems and instilling hope for recovery. In the middle sessions (2-9) participants will learn and practice interpersonal skills and offer and receive support from group members to resolve their problems. In the last session, they will review and celebrate progress and make plans to tackle future problems.
  Interventions: Behavioral: Interpersonal Psychotherapy Group
- Enhanced Usual Care (Active Comparator): Participants in the control arm will receive enhanced usual care. In intervention and control arms we will train health workers in health posts and primary care centres using the WHO mental health GAP Action training package. Participants in the control clusters will receive a handout with information about the location of these trained health workers and how they can access treatment. Participants in the control cluster reporting a current suicide plan or a suicide attempt in the past three months at baseline or in subsequent surveys will be assessed by a psychosocial counsellor employed through the project and offered one to one counselling as needed.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy Group — IPT is a psychological intervention that focuses on four common problems that trigger depression: grief, disputes, role transitions and social isolation. Using techniques and strategies such as linking mood to event and event to mood, role play and skill-building, IPT encourages the individual to analyse and improve their interpersonal relationships context. IPT was developed in the USA to treat depressed adults but it has also been used to treat other mental disorders and among different age groups.
  Arms: IPT-G
Behavioral: Enhanced Usual Care — Participants attending schools in the control arm will receive enhanced usual care. In intervention and control arms, we will train health workers in health posts and primary care centres using the WHO mental health GAP Action training package (mhGAP). Participants in the control clusters will receive a handout with information about the location of these trained health workers and how they can access treatment. Adolescents in the control cluster reporting a current suicide plan (i.e. in the past 2 weeks) or suicide attempt in the past three months will be assessed by a psychosocial counsellor employed through the project and offered counselling or referral to other services as per need.
  Arms: Enhanced Usual Care

SUMMARY:
Globally a third of adolescents are at risk of depression with negative consequences for their health and development. Most of the world's adolescents live in low- and middle-income countries (LMICs) where access to treatment for depression is limited. Psychological interventions are treatments that seek to change behaviours, cognitions and feelings to improve mental health but few have been tested with adolescents in LMICs. This study will use a cluster randomised controlled trial approach to test one such intervention, interpersonal therapy (IPT) for adolescents in Chitwan district, Nepal. The current study will compare whether adolescents (aged 13-18) with depression who receive group interpersonal therapy improve more than adolescents who receive information about local mental health services but no active intervention (enhanced usual care). Adolescents' depressive symptoms will be assessed eight to ten weeks after IPT has finished using the Patient Health Questionnaire modified for adolescents (PHQ-A). We will also aim to assess the feasibility and acceptability of delivering group IPT in secondary schools in Chitwan, Nepal. In addition, in this trial we aim to refine our hypotheses around why IPT works, how, and for whom, and pilot the tools which will be used to answer these questions later in the full trial.

DETAILED DESCRIPTION:
Depression and anxiety are leading causes of disability adjusted life years among adolescents aged 10-19 and can lead to social and educational impairment, substance misuse and suicide. The treatment gap for adolescent mental disorders is large, especially in low-and middle-income countries (LMICs). The WHO Mental Health Gap Action Programme outlines a role for psychological therapies in the treatment of child and adolescent emotional disorders such as depression and anxiety, however there is an urgent need to adapt these for use in LMICs. Between 2018 and 2020, our team including researchers and clinicians from TPO Nepal and King's College London adapted IPT for adolescents with depression in Nepal. Using an iterative mixed methods procedure, we adapted the WHO group IPT manual for delivery by school nurses and lay people in government secondary schools. We conducted an uncontrolled feasibility study of IPT with 62 adolescent boys and girls aged 13 to 19 in the mountainous district of Sindhupalchowk. Adolescents attended 82.3% (standard deviation 18.9) of group sessions. Depression and functional impairment improved between baseline and follow-up at 8-10 weeks post IPT: The Depression Self Rating Scale score decreased by 81% (95% confidence interval 70-95); functional impairment decreased by 288% (249-351).

Building on this previous research, we have designed a 4-stage, 5-year programme of work. The overall aim is to test the effectiveness and cost of scaling-up IPT in Nepal taking a "realist" evaluation approach where we will explore IPT's mechanisms of change and contextual factors that moderate its effects. This involves using formative research to develop an intervention theory of change from which we formulate hypotheses about how intervention mechanisms might interact with context to produce outcomes (context mechanism-outcome configurations, CMOCs).

According to this programme, Stage 1 (Formative Phase) is already completed. Currently we are applying for Stage 2, which is a pilot cluster randomized controlled trial (CRCT-pilot) of IPT for adolescent depression in Chitwan, a district in the lowland region of Nepal. As part of the current application, we aim to 1) test the feasibility and acceptability of the trial protocols, 2) pilot the qualitative and quantitative tools and 3) refine the theory of change hypotheses. Building on it, we will later apply for Stage 3 which will be a full cluster randomized controlled trial assessing the effectiveness/cost-effectiveness of IPT (CRCT-full) and Stage 4 which will consist of testing the CMOs using quantitative data from the full trial.

The study design is a parallel two-arm realist pilot cluster-randomised controlled trial. The trial will be conducted in eight schools (four intervention and four control). We will assess participants in intervention and control arms at baseline (week 0), after the second group session (week 4), after the sixth group session (week 8), at endline (weeks 13-14) and at follow-up (weeks 25-26). The acceptability of the intervention, randomisation, tools, uptake, utility of the intervention, facilitators' fidelity to the manual, mental health outcomes, and cost of design and delivery of the intervention will be assessed. The intervention process data will be also collected. This will include FGDs and interviews with adolescents and their parents, facilitators, nurses, teachers, and school principals to explore feasibility and acceptability of the intervention and study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Attending a participating school
* Enrolled in Class 8, 9 or 11
* Depressed (i.e. scoring 10 or more on the PHQ-A)
* Functionally impaired (i.e. scoring 4 or more on the functional impairment tool)

Exclusion Criteria:

* In Class 10 and 12 because these students will be busy preparing for School Education and Plus 2 exams
* In Class 7 because they may be too young to benefit from IPT
* Current suicide plan or attempted suicide in the past three months because these adolescents require more acute, intensive treatment
* Conversion disorder ("chhopne") in the past three months because group-based treatments may not be appropriate

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Depression | Baseline (week 0), after the second group session (week 4), after the sixth group session (week 8), at endline (weeks 13-14) and at follow-up (weeks 25-26)
  Patient Health Questionnaire for Adolescents (PHQ-A) will be used to measure depression. PHQ-A is a 9-item scale. It has a 4-point rating scale where 0 indicates 'not at all' and 3 indicates 'always'. The minimum scale score is 0 and the maximum is 27 with high score indicating severity of anxiety.

SECONDARY OUTCOMES:
Anxiety | Baseline (week 0), after the second group session (week 4), after the sixth group session (week 8), at endline (weeks 13-14) and at follow-up (weeks 25-26)
  Generalised Anxiety Disorder (GAD-7) will be used to measure anxiety. GAD-7 has 7-items and respondents are asked to score their experience of 7 common symptoms of anxiety in the past two weeks. It has a 4-point rating scale where 0 indicates 'not at all' and 3 indicates 'always'. The minimum scale score is 0 and the maximum is 21 with high score indicating severity of anxiety.
Functional Impairment | Baseline (week 0), after the second group session (week 4), after the sixth group session (week 8), at endline (weeks 13-14) and at follow-up (weeks 25-26)
  A locally-developed Functional impairment scale (FIS) will be used to measure impairment in daily activities. FIS is 11-item scale to assess impairment in daily functioning. It consists of 10-items, representing daily activities that adolescents generally do for themselves, family and community. It has a 4-point rating scale where 0 indicates "not at all' and 3 indicates "always". The total score of FIS ranges from 0 to 33 with higher score indicating more impairment in daily activities.
School Attendance | Baseline (week 0), after the second group session (week 4), after the sixth group session (week 8), at endline (weeks 13-14) and at follow-up (weeks 25-26)
  School attendance calculated as percentage of days attended in a standardised two-week period (excluding school closures).
PTSD | Baseline (week 0), after the second group session (week 4), after the sixth group session (week 8), at endline (weeks 13-14) and at follow-up (weeks 25-26)
  PTSD symptoms will be assessed with an 8-item shortened version of the PCL-5. It has a 4-point rating scale where 0 indicates "not at all' and 3 indicates "extremely". The total score ranges from 0 to 24 with higher score indicating more PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Gautam, MD, Study Director — Transcultural Psychosocial Organization Nepal

IPD SHARING:
Plan to Share IPD: Yes
The quantitative datasets generated during and/or analysed during the current study will be available upon request from Dr Kelly Rose-Clarke kelly.rose-clarke@kcl.ac.uk
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: The data is expected to be available when the data collection is complete. The expected date is June 2023.
Access Criteria: Individuals need to email Dr. Kelly Rose-Clarke (kelly.rose-clarke@kcl.ac.uk) with an intent statement explaining the purpose of the request